CLINICAL TRIAL: NCT05354622
Title: Investigating the Genetic Basis of Hereditary Spastic Paraplegia
Brief Title: Hereditary Spastic Paraplegia Genomic Sequencing Initiative (HSPseq)
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Boston Children's Hospital - Children's Rare Disease Cohorts Initiative (Unknown)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Principal Investigator, Boston Children's Hospital
Other Study IDs: P00039630
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Spastic Paraplegia; Neurodegenerative Diseases; Pediatric Disorder; Spasticity, Muscle; Motor Neuron Disease; Movement Disorders
Keywords: Hereditary Spastic Paraplegia; Neurodegenerative disease; Spasticity; SPG3a; SPG4; SPG11; SPG15; SPG26; SPG47; SPG50; SPG51; SPG52; Complex hereditary spastic paraplegia; Early Onset hereditary spastic paraplegia; Movement disorder; Adaptor protein complex 4; Neurogenetic disorder; Genetic Disease; Muscle Spasticity; Neurodevelopmental disorders; Musculoskeletal Disease
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Neurodegenerative Diseases; Muscle Spasticity; Motor Neuron Disease; Movement Disorders; Spastic paraplegia 3, autosomal dominant; Spastic paraplegia 26, autosomal recessive; Genetic Diseases, Inborn; Neurodevelopmental Disorders; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood sample or Buccal Swab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the HSP Sequencing Initiative is to better understand the role of genetics in hereditary spastic paraplegia (HSP) and related disorders. The HSPs are a group of more than 80 inherited neurological diseases that share the common feature of progressive spasticity. Collectively, the HSPs present the most common cause of inherited spasticity and associated disability, with a combined prevalence of 2-5 cases per 100,000 individuals worldwide.

In childhood-onset forms, initial symptoms are often non-specific and many children may not receive a diagnosis until progressive features are recognized, often leading to a significant diagnostic delay. Genetic testing in children with spastic paraplegia is not yet standard practice. In this study, the investigators hope to identify genetic factors related to HSP. By identifying different genetic factors, the investigators hope that over time we can develop better treatments for sub-categories of HSP based on cause.

DETAILED DESCRIPTION:
The hereditary spastic paraplegias (HSP) are a group of more than 80 inherited neurogenetic diseases that share the common feature of progressive spasticity. Collectively, the HSPs present the most common cause of inherited spasticity and associated disability, with a combined prevalence of 2-5 cases per 100,000 individuals worldwide. In childhood-onset forms, initial symptoms are often non-specific and many children may not receive a diagnosis until progressive features are recognized, often leading to a significant diagnostic delay. Genetic testing in children with spastic paraplegia is not yet standard practice.

The clinical diagnosis of HSP does not suggest anything about its molecular cause, with a wide range of outcomes dependent on the gene affected. The recent advances in HSP genetics speak to the importance of the field and the need for a more detailed study. Moreover, the relations between clinical features and genetic mechanisms are not well understood.

Given the influence of genetics on the likelihood of developing HSP as well as the complexity and diversity of the phenotypes, progress in HSP genetics will require efforts looking at relatively large samples of the HSP population. By bringing together very detailed phenotype information with high resolution DNA analyses, and using new approaches for comparing sequence information in candidate genes or looking for phenotype/genotype associations via genome-wide scanning, the investigators aim to be a leader in this emerging area of HSP research.

The aims of this study include:

1. To identify genetic findings (single nucleotide changes or copy number variants) in patients with progressive spastic paraplegia and related disorders.
2. To correlate molecular findings with HSP phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of progressive spasticity

Ages: 1 Month to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male or female, under 30 years, with suspected HSP
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2027-04-29 (Estimated); Study Completion 2027-04-29 (Estimated)

PRIMARY OUTCOMES:
Identify Genetic Findings | An average of 1 year
  Identifying genetic variants in patients with progressive spastic paraplegia
Correlating Genetic Findings with HSP Phenotypes | An average of 1 year
  Comparing phenotype/genotype associations via genome wide scanning

CONTACTS AND LOCATIONS:
Overall Officials: Darius Ebrahimi-Fakhari, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States